CLINICAL TRIAL: NCT05786313
Title: Prospective Controlled Clinical Study of Individualized, Precise and Standardized Posterior Cervical Open-door Surgery for Cervical Spinal Stenosis
Brief Title: Study of Individualized, Precise and Standardized Cervical Open-door Surgery for Cervical Spinal Stenosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: KY20222309-F-1
Record Dates: First submitted 2023-03-01; First posted 2023-03-27 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-02

CONDITIONS: Cervical Spinal Stenosis; Cervical Spinal Cord Injury; Individuation; Standardization
Keywords: cervical spinal stenosis; open angle

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Centerpiece titanium plate (Active Comparator): All surgical operations were performed by the same group of senior spine surgeons. The range of open door decompression involved C3 ~ C7. For convenient operation and more accurate statistics, the right side of the door axis and the left side of the door seam were selected for all operations. Centerpiece titanium plates were used for intraoperative fixation.
  Interventions: Procedure: Centerpiece titanium plate
- 3D printed arch titanium plate (Experimental): Before surgery, according to the imaging results, according to the effective imaging indicators screened in the early stage and the calculated door opening Angle formula, the door opening Angle of the patient's posterior cervical vertebra and the size of the fitted arch titanium plate were designed by mimics 10.0 software, and the titanium plate was printed using 3D printing technology. During the operation, the developed laminae opener was used to accurately control the door opening Angle and appropriate size titanium plate was installed for internal fixation. The standardized laminae door opening guide was used to complete the preparation of the door shaft side and door opening side of the lamina
  Interventions: Procedure: Centerpiece titanium plate

INTERVENTIONS:
Procedure: Centerpiece titanium plate — All indexes were collected from the patients with Centerpiece titanium plate for internal fixation.

SUMMARY:
To evaluate the safety and effectiveness of individualized, precise and standardized open-door posterior cervical surgery through a single-center, exploratory clinical study, so as to provide a more reliable basis for the treatment of cervical spinal stenosis.

ELIGIBILITY:
Inclusion Criteria:

* The age of 28-85 years old; Through systematic clinical and imaging examination, patients diagnosed with C3-7 multilevel cervical spondylitis myelopathy or cervical spinal stenosis who need to undergo posterior cervical open-door surgery.
* No contraindications in preoperative routine tests and examinations.
* Informed consent of patients.

Exclusion Criteria:

* Cervical radiculopathy
* Cervical kyphosis or instability
* Cervical spondylosis caused by trauma, tumor, tuberculosis and metabolic diseases
* Revision surgery or combined anterior-posterior surgery is required
* Serious neurological diseases affect the postoperative effect evaluation
* Mental illness cannot cooperate with follow-up
* Contraindications for MRI examination
* Patients themselves or their families do not agree to participate in the study
* Other situations that are not suitable for study participation.

Ages: 28 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
JOA score change | pre-operation,3 months after surgery, 6 months after surgery, 1 year after surgery
  Japanese Orthopedic Association (JOA) score is used to assess the function of spinal cord which is in the form of questionnaires. Postoperative improvement rate = ((postoperative score - preoperative score)/ (17- preoperative score)) X100%. Improvement rate can also correspond to the commonly used efficacy criteria: cure when the improvement rate is 100%, effective when the improvement rate is greater than 60%, effective when 25-60%, and ineffective when less than 25%.
NDI score change | pre-operation,3 months after surgery, 6 months after surgery, 1 year after surgery
  Neck Disability Index (NDI) score is used to assess the disorder of spinal cord which is in the form of questionnaires. Postoperative improvement rate = (total score)/ (numbers of program X5) X100%. Improvement rate can also correspond to the commonly used efficacy criteria: the improvement rate when 60%-80% means extremely severe dysfunction, when 40%-60% means severe dysfunction, when 20-40% means moderate dysfunction, and when less than 20% means mild dysfunction.
VAS score | pre-operation,3 months after surgery, 6 months after surgery, 1 year after surgery
  A Visual Analogue Scale (VAS) is used to measure the amount of pain that a patient feels ranges across a continuum from none to an extreme amount of pain. Using a ruler, the score is determined by measuring the distance (mm) on the 10cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.

SECONDARY OUTCOMES:
Maximum spinal cord compression change | pre-operation,3 months after surgery, 6 months after surgery, 1 year after surgery
  This index was measured by MRI, which was the ratio of the diameter of the cervical pulp at the most compressed segment to the mean diameter of the cervical pulp at the upper and lower segments without compression.
Compression ratio change | pre-operation,3 months after surgery, 6 months after surgery, 1 year after surgery
  This index was measured by MRI, which means the minimum sagittal diameter of the cervical pulp in the most compressed segment divided by maximum transverse diameter.
Transverse area change | pre-operation,3 months after surgery, 6 months after surgery, 1 year after surgery
  This index was measured by MRI, which means the cross-sectional area of the cervical pulp at the highest level of compression.

CONTACTS AND LOCATIONS:
Locations (1):
- Qi Wei, Xi'an, Shannxi Province, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmeiser G, Bergmann JI, Papavero L, Kothe R. Surgical Treatment of Multilevel Degenerative Cervical Myelopathy: Open-Door Laminoplasty and Fixation via Unilateral Approach. A Feasibility Study. J Neurol Surg A Cent Eur Neurosurg. 2022 Sep;83(5):494-501. doi: 10.1055/s-0041-1739224. Epub 2021 Dec 15. PMID 34911089
- [Background] Yeh KT, Lee RP, Chen IH, Yu TC, Liu KL, Peng CH, Wang JH, Wu WT. Laminoplasty instead of laminectomy as a decompression method in posterior instrumented fusion for degenerative cervical kyphosis with stenosis. J Orthop Surg Res. 2015 Sep 4;10:138. doi: 10.1186/s13018-015-0280-y. PMID 26338009
- [Background] Chen H, Liu H, Zou L, Li T, Gong Q, Song Y, Zeng J, Liu L, Kong Q. Effect of Mini-plate Fixation on Hinge Fracture and Bony Fusion in Unilateral Open-door Cervical Expansive Laminoplasty. Clin Spine Surg. 2016 Jul;29(6):E288-95. doi: 10.1097/BSD.0000000000000131. PMID 25023712
- [Background] Yuan W, Zhu Y, Liu X, Zhu H, Zhou X, Zhou R, Cui C, Li J. Postoperative three-dimensional cervical range of motion and neurological outcomes in patients with cervical ossification of the posterior longitudinal ligament: Cervical laminoplasty versus laminectomy with fusion. Clin Neurol Neurosurg. 2015 Jul;134:17-23. doi: 10.1016/j.clineuro.2015.04.004. Epub 2015 Apr 17. PMID 25929463